CLINICAL TRIAL: NCT06816628
Title: Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University
Brief Title: Effects of Comedy Therapy on Pain and Comfort Levels in Liver Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: okutan5
Record Dates: First submitted 2025-01-31; First posted 2025-02-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Liver Transplant; Complications; Pain, Postoperative; Care Acceptor, Health
Keywords: pain; comfort; transplant; liver; post-operatif
MeSH Terms: conditions — Pain, Postoperative; Patient Acceptance of Health Care; Pain

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pre-testpost- test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A patient introduction form, numerical rating scale and general comfort scale were applied as a pre-test after transplantation surgery. After patients came to the clinic after transplantation surgery and their condition was stable, 10-minute Turkish comedy films prepared by the researchers were shown. After the intervention, a numerical rating scale and general comfort scale were applied as a post-test. While patients watched the comedy films, a quiet and calm environment was provided in the patient room.
  Interventions: Other: comedy therapy
- Control Group (No Intervention): A patient introduction form, numerical rating scale and general comfort scale were applied as a pre-test after transplantation surgery. No intervention was made to the control group patients outside of the clinical protocol. After patients came to the clinic after liver transplantation and their condition was stable, the numerical rating scale and general comfort scale were applied again.

INTERVENTIONS:
Other: comedy therapy — After patients came to the clinic after transplantation surgery and their condition was stable, 10-minute Turkish comedy films prepared by the researchers were shown.
  Arms: Intervention Group

SUMMARY:
This study was conducted to investigate the effects of watching excerpts from classical Turkish comedy films on pain and comfort levels in liver transplant recipients during the postoperative period.

H1-0: Watching classical Turkish comedy films has no effect on postoperative pain in liver transplant recipients.

H1-1: Watching classical Turkish comedy films reduces postoperative pain in liver transplant recipients.

H2-0: Watching classical Turkish comedy films has no effect on postoperative comfort levels in liver transplant recipients.

H2-1: Watching classical Turkish comedy films increases postoperative comfort levels in liver transplant recipients.

DETAILED DESCRIPTION:
Intervention Group A patient introduction form, numerical rating scale and general comfort scale were applied as a pre-test after transplantation surgery. After patients came to the clinic after transplantation surgery and their condition was stable, 10-minute Turkish comedy films prepared by the researchers were shown. After the intervention, a numerical rating scale and general comfort scale were applied as a post-test. While patients watched the comedy films, a quiet and calm environment was provided in the patient room.

Control Group A patient introduction form, numerical rating scale and general comfort scale were applied as a pre-test after transplantation surgery. No intervention was made to the control group patients outside of the clinical protocol. After patients came to the clinic after liver transplantation and their condition was stable, the numerical rating scale and general comfort scale were applied again.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Being a liver transplant recipient,
* Data obtained after transplantation,
* Not having any visual or auditory problems.

Exclusion Criteria:

* Being under 18 years of age,
* Having any visual/auditory problems,
* Not accepting to participate in the study/wanting to leave,
* Not providing hemodynamic instability (sudden change in vital signs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
pain level | It will take approximately 5 minutes
  Patients' pain level will be measured with a "numerical rating scale". In the form, 0 points are evaluated as "no pain", 1-3 points as "mild pain", 4-6 points as "moderate pain", 7 and above points as "severe pain".
comfort level | It will take approximately 30 minutes
  General Comfort Scale:
  The general comfort scale was created by taking as a guide the taxonomic structure that includes three levels and four dimensions that constitute the theoretical components of comfort and is used to determine comfort requirements and to evaluate the situation of reaching the expected increase in comfort with nursing interventions that provide comfort. The scale is a four-point/six-point Likert type and contains a total of 48 items. The four-point Likert type was preferred in the study due to its ease of use. The lowest score that can be obtained from the scale is 48, the highest score is 192. High scores indicate a high level of comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, Dr., Principal Investigator — Study Principal Investigator Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)